CLINICAL TRIAL: NCT02278016
Title: Diagnosis Value of Procalcitonin, Interleukin-6, AgiotensininⅡin the Cerebrospinal Fluid of Patients With Central Nervous System Infective Diseases
Brief Title: Biological Markers for the Diagnosis of Central Nervous System Infective Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: xijing-120
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Infection
Keywords: procalcitonin; interleukin-6; agiotensininⅡ
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — procalcitonin,interleukin-6,agiotensininⅡ
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bacterial meningitis is a potentially life-threatening disease that is associated with substantial neurological morbidity and mortality. Accurate diagnosis is essential to improve outcome and prevent antibiotic overuse. Here we try to explore new biological markers for the diagnosis of the central nervous system infection disease.

DETAILED DESCRIPTION:
To investigate the diagnosis value of procalcitonin,interleukin-6, agiotensininⅡin the cerebrospinal fluid in the central nervous system infection disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 13 years or older;
2. At least two of the following clinical characteristics:headache, fever, neck stiffness, mental symptoms or consciousness impairment or seizures
3. Patients' family signed informed consent.

Exclusion Criteria:

1. Contraindications to lumbar puncture
2. Patients with active malignancy

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: More than 12 years old; meet the clinical diagnostic criteria for the central nervous system infection disease
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Levels of procalcitonin, interleukin-6, agiotensininⅡ in the serum and cerebrospinal fluid | 36 months
  meet the clinical diagnostic criteria for the central nervous system infection disease, the blood and cerebrospinal fluid samples after onset.

CONTACTS AND LOCATIONS:
Overall Officials: jiang wen, MD, Study Chair — The Department of Neurology , Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Li W, Sun X, Yuan F, Gao Q, Ma Y, Jiang Y, Yang X, Yang F, Ma L, Jiang W. Diagnostic Accuracy of Cerebrospinal Fluid Procalcitonin in Bacterial Meningitis Patients with Empiric Antibiotic Pretreatment. J Clin Microbiol. 2017 Apr;55(4):1193-1204. doi: 10.1128/JCM.02018-16. Epub 2017 Feb 8. PMID 28179405